CLINICAL TRIAL: NCT02054260
Title: Surgicel® (Fibrillar) in Non-variceal UGI Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Su Jin Hong, Professor, Soonchunhyang University Hospital
Other Study IDs: SCHBC_IRB_2013-40
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Non-variceal Upper Gastrointestinal Bleeding
MeSH Terms: interventions — Surgicel

ARMS (1):
- Surgicel add therapy (Experimental)
  Interventions: Drug: Surgicel

INTERVENTIONS:
Drug: Surgicel

SUMMARY:
The aim of this study is to assess of effect of Surgicel® (Fibrillar) for preventing delayed bleeding after endoscopic hemostasis in non-variceal upper gastrointestinal bleeding

ELIGIBILITY:
Inclusion Criteria:

* Patients with non variceal upper gastrointestinal bleeding proven by esophagogastroduodenoscopy
* Patients with active bleeding (Forrest classification Ia or Ib or IIa)

Exclusion Criteria:

* Patients with upper gastrointestinal tract malignancy
* Patients with acute severe illness
* Coagulopathy: liver cirrhosis, thrombocytopenia
* Pregnant women

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Rebleeding rate at the second look endoscopy | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Disease Center and Research Institute, Department of Internal Medicine, Soonchunhyang University College of Medicine, Bucheon-si, South Korea